CLINICAL TRIAL: NCT00979914
Title: Effect of an Education Programme for Patients With Osteoarthritis in Primary Care - a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Region Skåne, Primary health care, Sweden (Unknown)
Responsible Party: Principal Investigator, Eva Ekvall Hansson, Associate professor, Lund University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEPOA
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis in the Hip, Knee and Hand
Keywords: osteoarthritis; patient education; function; physio therapy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient education programme (Experimental): Patients with osteoarthritis who were referred to the patient education programme.The patients followed the patient education programme.
  Interventions: Other: Patient education programme
- Control (No Intervention): Patients randomized to control group

INTERVENTIONS:
Other: Patient education programme — The intervention consisted of five group sessions, three hours for each session. The focus was on self-efficacy. Eight to ten patients participated in the programme at the same time.
  Arms: Patient education programme

SUMMARY:
Osteoarthritis is a common disease. The core treatment is often patient education. The aim of this study is therefore to study the effect of a patient education programme for patients with osteoarthritis in primary health care.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a degenerative disease, considered to be one of the major national diseases that cause suffering for affected patients and costs for society.The predominant symptoms are pain, stiffness and impaired quality of life, often together with psychological distress. Treatment often consists of medication. Later in the disease, when the joint is destroyed, joint replacement surgery commonly occurs. Physical exercises aimed to increase muscle strength, endurance, proprioception and stability have proved to influence cartilage as well as function, symptoms and quality of life positively. Physical exercise may also reduce the need for hospital care after knee joint replacement.

Research suggests that patient education is feasible and valuable in terms of improvements in quality of life, in function, in well-being and improved coping . Accordingly, guidelines recommend education as a core treatment for osteoarthritis.

Patient education programmes are often defined as a planned learning experience to influence a patient's knowledge and health behaviour [13]. There are various types of patient education. It can be given by a physician as part of consultation, in small groups or delivered by a multi-disciplinary team [13, 14] Since 1994, Primary Health Care in Malmö has used a patient education programme directed towards OA. The programme has been developed by physiotherapists and occupational therapists in primary health care and has been implemented in the ordinary work.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of osteoarthritis

Exclusion Criteria:

* Must be able to speak and understand swedish

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
EQ5D | At baseline and at follow-up after 6 months
Arthritis self-efficacy scale | At baseline and at follow up after 6 months
One-leg rising from sitting to standing | At baseline and at follow up after 6 months
Grip Ability Test | At baseline and at follow up after 6 months

SECONDARY OUTCOMES:
Bipedal rising from sitting to standing | At baseline and at follow up after 6 months
One-legged jump | At baseline and at follow up after 6 months
Standing on one leg with eyes open and standing on one leg with eyes closed | At baseline and at follow up after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ekvall Hansson, PhD, Principal Investigator — Lund University
Locations (1):
- Primary Health Care, Malmo, Skåne County, Sweden

REFERENCES:
- [Background] Rosemann T, Joos S, Laux G, Gensichen J, Szecsenyi J. Case management of arthritis patients in primary care: a cluster-randomized controlled trial. Arthritis Rheum. 2007 Dec 15;57(8):1390-7. doi: 10.1002/art.23080. PMID 18050178
- [Background] Fransen M, Edmonds J. Reliability and validity of the EuroQol in patients with osteoarthritis of the knee. Rheumatology (Oxford). 1999 Sep;38(9):807-13. doi: 10.1093/rheumatology/38.9.807. PMID 10515639
- [Derived] Hansson EE, Jonsson-Lundgren M, Ronnheden AM, Sorensson E, Bjarnung A, Dahlberg LE. Effect of an education programme for patients with osteoarthritis in primary care--a randomized controlled trial. BMC Musculoskelet Disord. 2010 Oct 25;11:244. doi: 10.1186/1471-2474-11-244. PMID 20969809
- See also: Description of the EQ5D — http://www.euroqol.org/